CLINICAL TRIAL: NCT06715813
Title: Additional Effects of Transversus Abdominial Strengthening Along With Pelvic Floor Muscle Strengthening on Stress Urinary Incontinence Among Multiparous Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/54
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive SNAGs and the second will receive Sternocleidomastoid Release along with SNAGS. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic floor strengthening group (Active Comparator): Group A that is the control group will includes pelvic floor strengthening exercises. given three times a week on alternate days and session will be given for 4 weeks (protocol) and the retention effect will be given for 8 weeks. Each session will be performed at a moderate intensity , indicated by sustained contractions for 5 seconds initially and then progresively increased to 10 seconds overtime.
  pelvic floor strengtheing exercises includes :
  1. breathing exercises,
  2. kegels exercises
  3. bridging exercises
  4. squatting
  5. Elevator exercises
  Interventions: Procedure: pelvic floor strengthening
- PFMS + Transversus abdominal strengthening (Experimental): group B includes interventional group which includes core stabilization exercises for 2 weeks like stomach hallowing , dead bugs and pelvic tilt exercises and after 2 weeks dead bug progression, planks and pelvic floor strengthening exercises.
  Interventions: Procedure: pelvic floor strengthening; Procedure: Transversus abdominal strengthening

INTERVENTIONS:
Procedure: pelvic floor strengthening — pelvic floor strengthening exercises includes :
  1. breathing exercises,
  2. kegels exercises
  3. bridging exercises
  4. squatting
  5. Elevator exercises
Procedure: Transversus abdominal strengthening — core stabilization exercises for 2 weeks like stomach hallowing , dead bugs and pelvic tilt exercises and after 2 weeks dead bug progression, planks
  Arms: PFMS + Transversus abdominal strengthening

SUMMARY:
SUI stands for stress urinary incontinence. A common condition seen among multiparous women associated with physical strain like bending, coughing, sneezing that put strain on the pelvic floor muscles.

ELIGIBILITY:
Inclusion Criteria:

* Age group: multiparous women ( 30-50 yrs)
* females only
* all modes of delivery of childbirth
* diagnosed cases of SUI from fauji foundation hospital.
* patient without any medical contraindications and limitations (Sign and Symptoms of SUI)
* accordances with the michigan incontinence index

Exclusion Criteria:

* pregnancy or recent childbirth
* any history of pelvic organ prolapse or surgical intervention
* metabolic diseases, uncontrolled hypertension as well as neurological intervention
* any kind of malignancy in lower abdomen

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Age group: multiparous women ( 30-50 yrs)
Enrollment: 46 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
stress urinary incontinence | 8 weeks
  SUI will be measured using Michigan incontinence index

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan